CLINICAL TRIAL: NCT02131623
Title: Validation of the ItchRO Diaries in Pediatric Cholestatic Liver Disease
Brief Title: Validation of the Itch Reported Outcome (ItchRO) Diaries in Pediatric Cholestatic Liver Disease
Status: Completed | Type: Observational
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUM1038
Record Dates: First submitted 2014-05-01; First posted 2014-05-06 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Alagille Syndrome; Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Alagille Syndrome; Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Validation Group: Subjects with ALGS or PFIC and/or their caregivers

SUMMARY:
The purpose of the study is to validate the ItchRO instrument (a clinical outcome assessment measure of itching) prior to the analysis of longitudinal treatment effect data being generated in ongoing clinical trials.

DETAILED DESCRIPTION:
This research will examine the psychometric performance of the electronic diaries for the itch-reported outcome (ItchRO) measure for both patients and caregivers in a stand-alone 2-week validation study in the target patient population. The study is non-interventional in nature; the purpose of the study is to validate the ItchRO prior to the analysis of longitudinal treatment effect data being generated in ongoing clinical trials. Following training and initial completion of the electronic diaries, families will return home and complete the diaries twice daily over the course of two weeks. Additional assessments include the numerical rating scale to assess itching, the patient impression of change (PIC), the caregiver impression of change (CIC), PedsQL (pediatric quality of life), children's sleep habits questionnaire (CSHQ), and clinical scratch scale.

Longitudinal data will be used to follow the natural (non-interventional) course of the disease and the quality of the data. Test-retest reliability will be assessed using diary data from Day 1 to Day 14 in stable subjects as measured by the PIC for the child-completed measure and the CIC for the caregiver measure. Convergent validity (correlations between the ItchRO and similar concepts on the other measures included in the study) will also be explored (such as the correlation between sleep and morning ItchRO diary scores). Clinical validity (correlation between the ItchRO and clinician reports) and preliminary responsiveness of those who changed in their itching status over the two week period will also be assessed if sample sizes allow.

ELIGIBILITY:
Inclusion Criteria for subjects with ALGS or PFIC

1. The subject has voluntarily provided verbal assent or written assent in accordance with the site's Institutional Review Board (IRB) guidelines;
2. The subject's legal guardian has voluntarily provided permission for study participation and authorization for access to personal health information in conjunction with HIPPA;
3. The subject has a diagnosis of ALGS or PFIC;
4. The subject is able to speak and comprehend US English (applicable only for children age 5 and older);
5. The subject is willing and able to participate in the two-week validation study (applicable only for children age 5 and older); and
6. The subject is able to understand the nature, scope, and possible consequences of the study, and/or does not present evidence of an uncooperative attitude (applicable only for children age 5 and older).

Inclusion Criteria for caregivers of subjects with ALGS or PFIC:

1. The caregiver voluntarily provided written informed consent;
2. The caregiver is 18 years of age or older;
3. The caregiver has served as a consistent caregiver for the subject with ALGS or PFIC;
4. The caregiver's child or subject with ALGS or PFIC meets all of the study inclusion criteria for subjects with ALGS or PFIC;
5. The caregiver is able to speak, read, write, and comprehend US English;
6. The caregiver is willing and able to participate in the two-week validation study; and
7. The caregiver is able to understand the nature, scope, and possible consequences of the study, and/or does not present evidence of an uncooperative attitude.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects (children) with ALGS or PFIC and/or caregivers of subjects with ALGS or PFIC
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Validation of ItchRO measure | 2 weeks
  Validate the ItchRO measure with subjects with Alagille Syndrome (ALGS) or Progressive Familial Intrahepatic Cholestasis (PFIC) and/or their caregivers through the completion of the electronic diary twice daily over the course of two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Mirum
Locations (5):
- United States (4):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Children's Hospital Colorado, Aurora, Colorado
  - St. Louis Children's Hospital, St Louis, Missouri
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- The Hospital for Sick Children, Toronto, Ontario, Canada